CLINICAL TRIAL: NCT01194882
Title: Evaluation of Insuman Implantable 400 IU/ml in Patients With Type 1 Diabetes Treated With the Medtronic MiniMed Implantable Pump System Using Insuplant 400IU/ml
Brief Title: Benefit/Risk Evaluation of Insuman Implantable Versus Insuplant Using Medtronic MiniMed Implantable Pump System in Patients With Type 1 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUBIN_L_05335; 2010-021373-37 (EudraCT Number); U1111-1116-7658 (Other: UTN)
Record Dates: First submitted 2010-09-02; First posted 2010-09-03 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin; Metabolism

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Insuman Implantable (Experimental): Starting dose regimen is the same as the one administered to the patient prior randomization, then the insulin odse is established by the investigator on a patient basis in respect to the American Diabetes Association guidelines.
  Interventions: Drug: HUMAN INSULIN (BIOSYNTHETIC)
- Insuplant (Active Comparator): Starting dose regimen is the same as the one administered to the patient prior randomization, then the insulin odse is established by the investigator on a patient basis in respect to the American Diabetes Association guidelines.
  Interventions: Drug: Insuplant

INTERVENTIONS:
Drug: HUMAN INSULIN (BIOSYNTHETIC) — Pharmaceutical form: solution for infusion Route of administration: Intraperitoneal use Dose regimen: 400 IU/ml
  Other Names: HR1799
  Arms: Insuman Implantable
Drug: Insuplant — Pharmaceutical form:solution for infusion Route of administration: Intraperitoneal use
  Dose regimen:
  Other Names: Human insulin semi synthetic porcine derived
  Arms: Insuplant

SUMMARY:
Primary Objective:

To compare Insuman Implantable 400 IU/ml versus Insuplant 400 IU/ml with respect to the pump refill accuracy during a 4 refill cycle period (i.e. the comparative phase); To assess efficacy measured by hemoglobin glycosylated (HBA1c) change in Insuman Implantable 400 IU/ml group versus Insuplant 400 IU/ml group after a 4 refill cycle period (i.e. the comparative phase).

Secondary Objective:

To assess efficacy, safety, refill accuracy evolution and device interventions during the open-label treatment period with Insuman To evaluate daily insulin doses To assess Anti-Insulin Antibodies (ADAs or AIA) levels during all study phases

DETAILED DESCRIPTION:
The study duration will be displayed in 2 parts as follow:

Comparative phase (only French patients): 160 +/- 20 days Open label Insuman Implantable extension phase (French and European patients): from day 160 up to the grant of Insuman implantable marketing authorization

ELIGIBILITY:
Inclusion criteria:

1. Patients already treated with Insuplant 400 IU/ml via a Medtronic Implantable System 2007
2. Glycosylated hemoglobin ≤9.0%
3. Patient showing a percentage of error at refill equal or below 20%
4. Patient undergoing NaOH rinse procedure of at least 10 minutes period with or without flush Or Patient being re-implanted with a new pump (first fill with insulin)
5. Signed informed consent form prior to enrolment

Exclusion criteria:

1. Pump life time > 6 years
2. Pump battery voltage < 2.6 volts
3. Pregnancy or childbearing potential without a medically approved form of birth control

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 479 (Actual)
Dates: Start 2010-11-16; Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Refill accuracy between the 2 insulin groups | During 4 refill cycles
Change in glycosylated hemoglobin (HbA1c) | From baseline to 6 months

SECONDARY OUTCOMES:
Occurrence of Hypoglycaemia (asymptomatic and symptomatic hypoglycaemia, severe and serious symptomatic hypoglycaemia | From baseline to 6 months
Occurrence of hyperglycaemia | From baseline to 6 months
Occurrence of diabetic ketoacidosis | From baseline to 6 months
Change in insulin dose | From baseline to 6 months
Antibody assessments (anti-Insulin antibodies) | From baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (17):
- Investigational Site Number 056-001, Leuven, Belgium
- France (12):
  - Investigational Site Number 250-004, Corbeil-Essonnes
  - Investigational Site Number 250-008, Dijon
  - Investigational Site Number 250-003, Dommartin-lès-Toul
  - Investigational Site Number 250-012, Le Mans
  - Investigational Site Number 250-009, Lille
  - Investigational Site Number 250-007, Marseille
  - Investigational Site Number 250-001, Montpellier
  - Investigational Site Number 250-005, Paris
  - Investigational Site Number 250-010, Pessac
  - Investigational Site Number 250-011, Saint-Priest-en-Jarez
  - Investigational Site Number 250-002, Strasbourg
  - Investigational Site Number 250-006, Toulouse
- Netherlands (3):
  - Investigational Site Number 528002, Roermond
  - Investigational Site Number 528003, The Hague
  - Investigational Site Number 528001, Zwolle
- Investigational Site Number 752-001, Stockholm, Sweden

REFERENCES:
- [Derived] Schaepelynck P, Riveline JP, Renard E, Hanaire H, Guerci B, Baillot-Rudoni S, Sola-Gazagnes A, Catargi B, Fontaine P, Millot L, Martin JF, Tachouaft H, Jeandidier N; EVADIAC Group. Assessment of a new insulin preparation for implanted pumps used in the treatment of type 1 diabetes. Diabetes Technol Ther. 2014 Sep;16(9):582-9. doi: 10.1089/dia.2013.0369. Epub 2014 Apr 15. PMID 24735100